CLINICAL TRIAL: NCT05805930
Title: Therapeutic Approach in Colchicine-resistant Recurrent pEricarditis in Children: an Open-label Randomized Trial Comparing Anakinra vs sTEroids
Brief Title: Therapeutic Approach in Colchicine-resistant Recurrent pEricarditis in Children
Acronym: CREATE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Istituto Giannina Gaslini (Other)
Responsible Party: Principal Investigator, Nicolino Ruperto, MD, MPH, Head of Trial Centre, Istituto Giannina Gaslini
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREATE
Record Dates: First submitted 2023-03-23; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Pericarditis
MeSH Terms: conditions — Pericarditis | interventions — Interleukin 1 Receptor Antagonist Protein; Prednisone; Steroids; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Steroids (Active Comparator): Treatment with prednisone will be initiated at a dosage of 1 mg/kg/day (maximum 50 mg/day) in twice daily administration for 14 days. In case of complete response to treatment, prednisone will be reduced from day 14, otherwise it will be continued at 1 mg/kg/day until day 28 (week 4). Patients with complete response at day 28 will continue the study entering part 2, in which therapy will be progressively tapered.
  In part 2, prednisone will be tapered progressively by 0.1-0.15 mg/kg/day of prednisone (or 5 mg in patients on the maximum dose of 50 mg/day) from current treatment every week until the break. If there is no relapse, treatment will be discontinued over a 10-week period. Patients will then be evaluated every 4 weeks until the end of the study (week 24).
  Interventions: Drug: Prednisone
- Arm 2: Anakinra (Experimental): Treatment with anakinra will be initiated at a dose of 2 mg/kg/day (maximum dose 100 mg/day) as a single daily dose and maintained until day 28 (week 4).
  Patients who achieve a complete treatment response at week 4 (day 28) will continue the study into Part 2. Patients without a complete treatment response will drop out of the study.
  In Part 2 patients will continue daily anakinra treatment through week 12. The treatment will then be progressively reduced through the reduction of one weekly administration of the drug. The reductions will be made every 2 weeks until the interruption. Therefore, if no relapse occurs, treatment will be discontinued at week 24.
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — : Patients will continue daily treatment with anakinra up to week 12. Treatment will be then progressively tapered through the reduction of an administration of the drug per week. Reductions will be performed every 2 weeks up to discontinuation. Therefore, if a relapse does not occur, the treatment will be withdrawn at week 24.
  Arms: Arm 2: Anakinra
Drug: Prednisone — Steroids will be progressively tapered with a reduction of 0,1-0,15 mg/kg/day of prednisone (or 5 mg in patients in treatment with the maximum dosage of 50 mg/day) from the ongoing treatment every week up to discontinuation. If a relapse does not occur, the treatment will be withdrawn in a period of time of 10 weeks.
  Other Names: Steroid; Corticosteroid
  Arms: Arm 1: Steroids

SUMMARY:
The purpose of this study is to demonstrate that anakinra provides more rapid disease control than steroids in the first month of treatment in the event of recurrent pericarditis and is more effective in preventing further exacerbations in patients aged between eight months and eighteen years of age with idiopathic or post-procedural pericarditis, unresponsive to first-line treatment with NSAIDs and colchicine at the appropriate dosage, or in case of colchicine intolerance. The efficacy of the two treatments will be evaluated by the capacity and timing of the two therapies to determine a complete control (clinical, laboratory and instrumental) of the disease and the absence of recurrences.

DETAILED DESCRIPTION:
Although steroids represent the second-line treatment for recurrent pericarditis (RP), to be used in case of inadequate response to NSAIDs and colchicine, their use is controversial due to their side effects.

Indeed, in adult patients with RP it has been demonstrated that the use of steroids is associated with an increased risk of recurrence: in a study carried out in adult patients, 64% of patients taking high-dose steroids (> 1 mg/kg/ of prednisone or equivalent), and 32% of patients taking this low-dose drug (< 1 mg/kg/day of prednisone or equivalent) relapsed. Furthermore, the therapy is associated with serious side effects and an increased risk of hospitalization, especially in patients treated with high doses. Finally, a high percentage of RP patients (both adult and pediatric) treated with steroids tend to become steroid-dependent, experiencing a disease exacerbation during tapering of treatment or soon after its discontinuation. The side effects associated with the chronic use of steroids are well known, especially in childhood, as their use is associated not only with reduced bone density, but also with growth retardation. Therefore, their long-term use is contraindicated, especially in children.

In a recent retrospective study of 58 pediatric patients with recurrent pericarditis treated with IL-1 inhibitors, a high steroid dependence rate was observed (45 of 48 treated patients). In this study, the presence of predictive factors associated with the possibility of achieving long-term remission was evaluated. Unfortunately, it could not be shown that avoiding steroid use was associated with an increased chance of withdrawing anakinra without relapse. This is likely due to the large variability of the cohort included in the retrospective study.

Therapy with anakinra in recurrent pericarditis is aimed at obtaining rapid and complete control of the disease and maintaining it over time, allowing the suspension of steroid therapy and thus reducing the risk of complications, chronicity and recurrence.

In the field of pediatric rheumatology, there is convincing evidence that in children with chronic arthritis a more aggressive therapy at an early stage can take advantage of the so-called "window of opportunity": according to this theory, early biological treatment can modify the pathogenetic mechanism of the disease by improving its long-term outcomes.

In particular, it has been shown that anakinra therapy in children with systemic JIA can lead to rapid attainment of inactive disease and allow for early discontinuation of treatment in the absence of recurrence in the majority of patients. Among all the rheumatological pathologies of the pediatric age, systemic JIA is the one that has the greatest similarities with autoinflammatory diseases due to the presence of fever, sometimes recurrent, rash and serositis, typical characteristics of AID, especially of inflammasomopathies. Recurrent pericarditis itself has many similarities to these conditions, as demonstrated by the efficacy of interleukin-1 inhibition. In fact, both of these conditions are considered by many to be real autoinflammatory diseases, with a multifactorial etiology. It is therefore reasonable to think that the concept of the "window of opportunity" can also be translated to recurrent pericarditis: the early blockade of cytokines could in fact abrogate the pathogenetic mechanism of the disease and therefore its chronic course and/or its relapses.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients.
2. Parent or legal guardian written informed consent and child assent, if appropriate, are required before any assessment is performed.
3. Diagnosis of relapse of pericarditis in a patient with previous diagnosis of acute pericarditis (idiopathic or secondary to invasive cardiac procedures).
4. Inadequate response or intolerance to non-steroidal anti-inflammatory drugs or colchicine

Exclusion Criteria:

1. Pericarditis secondary to a known infection (viral, bacterial, mycobacterial).
2. Pericarditis in a patient with a previous diagnosis of any neoplasm and without complete recovery from at least one year.
3. Pericarditis in the context of a systemic disease.

   1. Patients fulfilling diagnostic criteria for an autoimmune systemic disease
   2. Patients with a previous diagnosis of a genetically confirmed autoinflammatory disease
4. Any conditions or significant medical problems, which in the opinion of the investigator places the patient at unacceptable risk for immunomodulatory therapy.
5. Main alteration in the blood count
6. Presence of Human Immunodeficiency Virus (HIV) infection, Hepatitis B or Hepatitis C infections.
7. Evidence of active or latent tuberculosis (TB) determined by positive QuantiFERON (QFT-TB G In-Tube) test or positive Purified Protein Derivative (PPD) test (≥5 mm induration) within 2 months prior to randomization.
8. Administration of any investigational drug or implantation of investigational device, or participation in another trial, within 30 days before screening.
9. Use of steroids at the dosage of 1 mg/kg/day of prednisone or equivalent for at least 5 days in the 30 days before randomization.
10. Live vaccinations within 1 months prior to the start of the trial and during the trial.
11. Pregnancy, confirmed by a positive hCG laboratory test.
12. Female adolescents (≤18 years of age) of childbearing potential who do not agree to abstinence or, if sexually active, do not agree to the use of contraception.

    -

Ages: 8 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with complete response to treatment | Day 7
  Complete response to treatment at day 7
Number of participants with disease Flare | 3 months
  Absence of flare after 3 months of therapy

SECONDARY OUTCOMES:
Time to response | Up to 24 weeks
  Time to respond to treatment
Number of participants with improved Quality of life | Up to 24 weeks
  Evaluation of quality of life through specific questionnaire

IPD SHARING:
Plan to Share IPD: No